CLINICAL TRIAL: NCT06227273
Title: Hydrogen Water Dosing Study for ME/CFS and Chronic Fatigue
Brief Title: Hydrogen Water Dosing Study for ME/CFS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Collaborators: Natural Wellness Now Health Products (Unknown)
Responsible Party: Principal Investigator, Fred Friedberg, Principal Investigator, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 41245
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Water

STUDY DESIGN:
Intervention Model Description: Two different 16-week dosing schedules will be compared: A standard dose of hydrogen water as compared to a standard dose followed by an increased dose of hydrogen water.
Who Masked: Investigator
Masking Description: The investigator is blinded to computer-generated condition assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H2 Standard Dose (Active Comparator): This condition will schedule 1-5 glasses of hydrogen water a day for 16 weeks.
  Interventions: Dietary Supplement: Hydrogen water
- H2 Standard Dose followed by Higher Dose H2 (Active Comparator): This condition will schedule 1-5 glasses of hydrogen water a day for 8 weeks followed by 4-5 glasses of hydrogen water for 8 weeks.
  Interventions: Dietary Supplement: Hydrogen water

INTERVENTIONS:
Dietary Supplement: Hydrogen water — Daily consumption of hydrogen water for 16 weeks.

SUMMARY:
The aim of this 16-week pilot randomized trial is to explore the potential benefit of the OTC supplement hydrogen water, for the symptoms of chronic fatigue syndrome (CFS). Methods: This 16-week home-based trial will compare two groups: (1) low dose hydrogen water (2-3 glasses/day) for all 16 weeks; and (2) low dose followed by high dose hydrogen water (up to 5 glasses/day). Condition (2) involves an initial 8 weeks of low dose H2 followed by 8 weeks of high dose H2 in order to test the premise that the higher dosage will be more effective with fewer adverse effects if preceded by several weeks of low dose H2. Outcomes measures will include online assessments of fatigue, physical function and stress. A salivary biomarker for oxidative stress, Uric Acid, will also be assessed.

DETAILED DESCRIPTION:
Previous clinical studies (8-12 week intervention trials) have indicated that H2 enriched water reduces concentrations of markers of oxidative stress in patients with metabolic syndrome, improves lipid and glucose metabolism in patients with type 2 diabetes, improves mitochondrial dysfunction in patients with mitochondrial myopathies, and reduces inflammatory processes in patients with polymyositis/ dermatomyositis (Mizuno et al., 2017). In addition to its potential therapeutic properties, H2 water is portable, easily administered and safe to ingest (Nagata et al., 2013). Owing to its potential therapeutic efficacy and lack of adverse effects, H2 may show promise for clinical use in ME/CFS. Two CFS studies conducted in the PI's laboratory (Friedberg and Choi, 2022; Friedberg and Choi, under review) yielded mixed findings. The initial randomized controlled trial showed no benefit for H2 water, but the second study, a randomized trial of H2 and heart rhythm biofeedback that was of longer duration (60 days) with a lower dosage of H2 water found significant improvements in fatigue and physical function. The new proposed randomized trial will extend treatment to 120 days and test a standard dosage of H2 water for all 120 days in group1 in comparison to standard dosage for the initial 60 days followed by increased dosage for the remaining 60 days (Group 2). Group 2 is may show a greater treatment effect once subjects are acclimated to the lower initial dose. Thus, we are testing different dosing schedules to determine which may be more effective in CFS.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 18-65 of both sexes; considered physically capable and willing to perform the study tasks.

* Meeting validated phone-screen eligibility for ME/CFS criteria.
* Patient has internet and computer.

Exclusion Criteria:

Cases of fatigue clearly attributable to self-report medical conditions such as untreated hypothyroidism, unstable diabetes mellitus, organ failure, chronic infections, and chronic inflammatory diseases, or AIDS.

__ Exclusionary psychiatric disorders include any psychosis, or alcohol/ substance abuse within two years prior to illness onset and any time afterward, and current or past depression with melancholic or psychotic features within 5 years prior to onset of ME/CFS or anytime afterward

* Pregnancy is an exclusion.
* Patients with BMI>35.
* Patients at significant risk of suicide or in need of urgent psychiatric treatment. As much as possible, appropriate medical and psychiatric referrals to facilities local to subjects will be provided.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 16 weeks
  Self-report measure of effect of fatigue on functioning.

SECONDARY OUTCOMES:
SF-36 PF | 16 weeks
  Self-report physical function measure
Depression, Anxiety and Stress Scale | 16 weeks
  Self-report measure of depression, anxiety and stress symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Fred Friedberg, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided